CLINICAL TRIAL: NCT03560648
Title: Innovative Device for the Evaluation of the "Motor Functional Age": How Old is Your Muscle?
Brief Title: Device Evaluating the Muscular Functional Age
Acronym: CHRONOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Université de Technologie de Compiegne (Other); Sorbonne University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: K170916J; 2018-A00909-46 (Other: IDCRB)
Record Dates: First submitted 2018-05-18; First posted 2018-06-18 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers; Skeletal Muscle
Keywords: muscle aging; sarcopenia; neuromuscular dysfunction
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reference group (Other): To define the normal muscle aging from HD-sEMG and accelerometer signals correlated to muscular parameters obtained from Dual Energy X-ray Absorptiometry (DEXA), handgrip strength and muscular echography. Data will be collected in healthy volunteers, aged 25 to 75 years old, physically active on IPAQ questionnaire.
  Interventions: Device: High definition surface electromyography combined with accelerometer
- Test group (Other): To evaluate the capacity of MFA to detect early muscle aging in " tests " individuals, sedentary volunteers within the same age group (45-55 years old).
  Interventions: Device: High definition surface electromyography combined with accelerometer

INTERVENTIONS:
Device: High definition surface electromyography combined with accelerometer — HD-sEMG and accelerometer data will be collected by Mobita 32® (TMSi) device.

SUMMARY:
The CHRONOS project aims to provide a device to detect earlier the motor decline, by developing a precise quantitative device measuring "Motor Functional Age" (MFA) of young, middle-aged and old people, thus preventing future functional motor loss for healthy aging. The MFA might be different from the Chronological Age (CA), depending on lifestyle, physical activity, and medical condition. Thus, this device will permit monitoring, adaptation and new design of a variety of personalized therapies for healthy aging including physical exercise, medication and nutritional interventions to reduce the MFA toward or less than the CA. The device combines data processing software that estimates the MFA by assessing muscle aging using a non-invasive multichannel electromyographical technique coupled to accelerometry sensors for motion evaluation. These data will provide with a built-in clinical database of subjects from different age categories (25-75 years old).

DETAILED DESCRIPTION:
Background:

Aging is accompanied by sarcopenia, defined by a loss in muscle mass (starting from the age of 25) and strength/function, leading to a decline in mobility. This functional motor decline is an increasing health problem with impairing functional independence and quality of life among seniors. Furthermore, a sedentary lifestyle reinforced by an abusive use of modern technology (videogames, transportation and communication) and poor dietary habits (often rich in sugar and fats and poor in high quality proteins) are more common in younger demographics than ever before. These unhealthy habits lead to premature muscle aging, sarcopenia and future functional motor loss.

Methods to easily and rapidly assess muscle quality in multiple clinical settings and with minimal patient burden are needed.

Moreover, an individual's CA, taken solely, is rarely a reliable index of an individual's ability to perform specific physical task. The proposed MFA concept is innovative since it precisely expresses the motor abilities through a sensitive screening of muscle activation using a recent HD-sEMG (High density-surface electromyogram) technique that is, by far, more robust, precise and representative than the classical single bipolar technique.

Aim and Objectives:

In the CHRONOS project, a device using HD-sEMG technology actually devoted to research actions only, even though CE-certified, will be designed by testing and combining data allowing one to assess the muscle activation efficiency and motion capacity (accelerometry sensors), as a function of CA.

* Main objective : attribute a MFA to define the normal muscle aging from HD-sEMG and accelerometer signals correlated to muscular parameters obtained from Dual Energy X-ray Absorptiometry (DEXA), handgrip strength and muscular echography. Data will be collected in " reference " individuals, healthy volunteers, aged 25 to 75 years old.
* Secondary objectives :

  1. to evaluate the capacity of MFA to detect early muscle aging in " tests " individuals, sedentary volunteers within the same age group (45-55 years old).
  2. study correlation between HD-sEMG/accelerometer signals and muscular parameters from DEXA, handgrip strength, physical performance by SPPB (Short Physical Performance battery), walking speed, walking distance in 6min, physical activity evaluated objectively by actimeter, and subjectively by IPAQ (International Physical Activity Questionnaire), muscle echography parameters, and nutritional data.

ELIGIBILITY:
Main inclusion criteria

* walking without help
* physically active (IPAQ questionnaire: moderately or highly active) for "reference group" and sedentary (IPAQ questionnaire: low activity) for "test" group.

Main exclusion Criteria

* Body mass index <18.5 and >= 30 kg/m2
* Neurological, endocrinological, rheumatologic, myopathy, orthopedic and severe cardio-respiratory diseases
* Non smoking and non alcoholism,
* Taking medications interfering with muscle function
* Pregnant

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Motor functional age determined by HD-sEMG (rectus femoris) during sit to stand | Day 0
  HD-sEMG data will be correlated to Skeletal Mass Muscle Index, handgrip strength and muscle echography data.
Motor functional age determined accelerometer signals during sit to stand | Day 0
  Accelerometer data will be correlated to Skeletal Mass Muscle Index, handgrip strength and muscle echography data.

SECONDARY OUTCOMES:
Skeletal Mass Muscle Index | Day 0
  Dual-energy x-ray absorptiometry (DEXA) is the imaging technique recommended for the diagnosis of sarcopenia. It gives minimal irradiation and gives an adequate estimate of the appendicular muscle mass (ALM). By dividing the ALM by the size in centimeters, we obtain the Skeletal Mass Muscle Index (SMI). SMI values below 2 standard deviations from the mean point towards sarcopenia.
Hand grip strength | Day 0
  By placing a dynamometer in the patient's hand and asking him to apply maximum pressure to it, the muscular strength of the extremities of the limbs is estimated.
Walking speed | Day 0
  Walking speed evaluates the muscular performance. The seated patient must walk a distance of 4 meters as quickly as possible without the help of a third party. It has been shown that there is a non-linear relationship between walking speed and muscle strength.
Short Physical Performance Battery (SPPB) | Day 0
  A battery of tests combining walking speed on 4 meters, sit-to-stand test and tandem balance test giving a physical performance score
Bone mineral density (T-score) | Day 0
  Dual-energy x-ray absorptiometry (DEXA) is the imaging technique recommended for bone mineral density measure
Muscle echography | Day 0
Walking distance in 6 minutes | Day 0
  Walking speed and distance evaluates the muscular performance. The seated patient must walk during 6minutes as quickly as possible without the help of a third party.
International Physical Activity Questionnaire (IPAQ) score | Day 0
  IPAQ assesses physical activity undertaken across a comprehensive set of domains including:a. leisure time physical activity; b. domestic and gardening (yard) activities; c. work-related physical activity; d. transport-related physical activity. Two types of scoring: continuous score (sum of MET-minutes/week, reflecting the intensity of physical activity) and categorical score (low/moderate/high level of physical activity) with criteria based on MET-minutes/week and type of reported physical activity (moderate, vigorous intensities).
Time to perform 5 sit-to-stand | Day 0
  Time in seconds
Physical activity | Day 7
  Physical activity assessed objectively by actimetry during 1 week
Sleep-wake duration | Day 7
  Sleep-wake duration assessed objectively by actimetry during 1 week
Sarcopenia stage | Day 0
  The sarcopenia stage will be assessed according to the European Working Group on Sarcopenia in Older People (EWGSOP) definition: "non sarcopenia", "pre-sarcopenia" and "sarcopenia"

CONTACTS AND LOCATIONS:
Overall Officials: Kiyoka KINUGAWA, MD, PhD, Principal Investigator — Charles Foix Hospital
Locations (1):
- APHP - Charles Foix Hospital, Ivry-sur-Seine, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Imrani L, Boudaoud S, Lahaye C, Moreau C, Ghezal M, Ben Manaa S, Doulazmi M, Laforet J, Marin F, Kinugawa K. High-density Surface Electromyography as Biomarker of Muscle Aging. J Gerontol A Biol Sci Med Sci. 2023 Jan 26;78(1):25-33. doi: 10.1093/gerona/glac143. PMID 35876634